CLINICAL TRIAL: NCT04227132
Title: Modulation of Visuospatial Awareness During Multi-tasking in Right Hemisphere Stroke Patients: Towards Novel Behavioural and Neurofunctional Predictors of Impairments and Recovery of the Attentional Networks
Brief Title: Evaluation of an Adaptive Computerized Training for Rehabilitation of Spatial Neglect in Stroke Survivors
Acronym: MULTITASK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Marco Zorzi, Professor, University of Padova
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RF-2013-02359306
Record Dates: First submitted 2019-12-31; First posted 2020-01-13 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Spatial Neglect; Neglect, Hemispatial; Attention Impaired; Cerebrovascular Disorders
Keywords: Neglect; Recovery of function; Rehabilitation; Videogame; Post-stroke
MeSH Terms: conditions — Stroke; Perceptual Disorders; Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: Both experimental and control trainings will be administered consecutively to all patients. Each type of training will be delivered for 10 sessions, with order of training randomized across participants.
Masking Description: Patients will be informed to take part in an experimental study on the rehabilitation of attention delivered through a computer game. Specific information about the rationale of the study will not be conveyed to patients. Both trainings will be administered, with the aim to support patients' autonomy in performance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labyrinth training, then Standard training (Experimental): Patients will receive at first the Labyrinth training for 10 sessions of 45 minutes, delivered 4 days per week. The, they will undergo the Standard training for 10 sessions of 45 minutes, for around 4 days per week. Before and after each training patients are tested for primary and secondary outcomes with standardized tests.
  Interventions: Device: Adaptive computer game training
- Standard training, then Labyrinth training (Experimental): Patients will receive at first the Standard training for 10 sessions of 45 minutes, delivered 4 days per week. Then they will undergo the Labyrinth training for 10 sessions of 45 minutes, for around 4 days per week. Before and after each training patients are tested for primary and secondary outcomes with standardized tests.
  Interventions: Device: Standard computerized training

INTERVENTIONS:
Device: Adaptive computer game training — Patients sit in front of a computer monitor and play the adaptive videogame with a joystick. The game requires to orient and move inside a maze, and it includes phases that engage multitasking abilities. The level and speed of the game is adapted online to patients' performance.
  Arms: Labyrinth training, then Standard training
Device: Standard computerized training — Patients sit in front of the computer monitor and perform simple computerized exercises using a keyboard to respond. Exercises are organized into modules according to the trained cognitive functions. Patients will perform four different modules that are designed for neglect rehabilitation. The level of exercises adapts periodically based on patient's performance.
  Arms: Standard training, then Labyrinth training

SUMMARY:
The aim of this study is to investigate the effect of training with an adaptive computer game, in comparison to standard training, in the rehabilitation of stroke survivors suffering from spatial neglect.

DETAILED DESCRIPTION:
Many stroke survivors who have suffered right brain damage show spatial neglect (SN), a deficit of spatial attention orienting that causes unawareness for stimuli located in the left hemispace. Recent data show that the execution of concurrent tasks (that is, multitasking) can worsen the clinical condition and impact functional recovery.

The aim of this study is to investigate the effect of an adaptive computer game "Labyrinth" previously validated on health population. The videogame is designed for training both attention and execution functions as it engages spatial navigation and multitasking. The effect of the computer game will be compared to standard computerized exercises used for neglect rehabilitation.

The investigators plan to administer to a sample of 30 stroke patients with SN both Labyrinth and standard trainings for 10 sessions each. The two trainings will be delivered in a randomized crossover design. Improvements of patients' performance will be registered across trainings and in a follow-up test at 1 month, by assessing the severity of SN and functional everyday outcomes. The investigators expect that patients' performance will improve following both types of training, but with stronger improvement for the adaptive videogame.

ELIGIBILITY:
Inclusion Criteria:

* First stroke patients with right brain damage
* Right-handed
* Preserved Italian language comprehension to provide informed consensus
* Clinical signs of spatial neglect (diagnosis by BIT)

Exclusion Criteria:

* Prior history of psychiatric or neurological disease
* Substance abuse
* Inability to sustain the experimental trainings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes at Behavioral Inattention Test (BIT) | Baseline; immediately after the first training; immediately after the second training; finally after 3 weeks from the end of second training
  Diagnostic test for spatial neglect, composed by different subtests of spatial attention
Changes at KF-NAP scale | Baseline; immediately after the first training; immediately after the second training; finally after 3 weeks from the end of second training
  Test for everyday functional outcome

SECONDARY OUTCOMES:
Changes at Load Test | Baseline; immediately after the first training; immediately after the second training; finally after 3 weeks from the end of second training
  Computerized test on spatial monitoring and multitasking abilities
Changes at Apple Test | Baseline; immediately after the first training; immediately after the second training; finally after 3 weeks from the end of second training
  Test for allocentric and egocentric spatial neglect

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zorzi, Ph.D., Principal Investigator — Department of General Psychology, University of Padua, Padua, Italy
Locations (1):
- Ospedale San Camillo IRCCS, Venice-Lido, Veneto, Italy

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963